CLINICAL TRIAL: NCT02909998
Title: Evaluation of Predictive Genetic Markers of Response to Biologic Therapies in Chronic Arthritis
Brief Title: Biomarkers in Chronic Arthritis
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8359; 2008-A01087-48 (Other: FRANCE: Agence française de Sécurité Sanitaire des Produits de Santé)
Record Dates: First submitted 2016-09-08; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Arthritis
Keywords: Biomarkers; Genetic; Chronic arthritis; Treatment
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood sample — Conservation at the end of the blood sample

SUMMARY:
Use of genotyping for the optimization of treatment with biologics in chronic arthritis by looking for an association between certain alleles and response to treatment.

DETAILED DESCRIPTION:
Chronic arthritis in children and in adults represent a public health problem in number and difficulty of treatment. 30% of patients are non-responders and / or relapse upon discontinuation of treatment. Some of these treatments are not always well tolerated, sometimes with infectious complications including tuberculosis limiting the use of biological therapies. This study will validate a battery of genetic markers to predict responders biotherapy, determine the prognosis of patients, these treatments are reserved for the most severe forms, and thus improve the care of patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with biotherapy may be included in this study with all information necessary for regular medical consultations (filling specific monitoring by GPs questionnaires), physical therapists visits, occupational therapists, psychologists.. etc

Exclusion Criteria:

* Patients treated with biological therapy for non rheumatic disease
* Other inflammatory diseases such as Crohn's disease
* Refusal to participate in the collection

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients referred for chronic arthritis
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2008-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of responsive patients with a given polymorphism (%) | At the inclusion

SECONDARY OUTCOMES:
Distribution of patients with a given biotherapy (%) | At the inclusion
Distribution of patients presenting a given polymorphism (%) | At the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle TOUITOU, MD, PhD, Principal Investigator — Montpellier Hospital University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ladhari C, Le Blay P, Vincent T, Larbi A, Rubenstein E, Lopez RF, Jorgensen C, Pers YM. Successful long-term remission through tapering tocilizumab infusions: a single-center prospective study. BMC Rheumatol. 2020 Feb 28;4:5. doi: 10.1186/s41927-019-0109-0. eCollection 2020. PMID 32161846